CLINICAL TRIAL: NCT06719271
Title: Postural Stability of Ambulatory Children With Cerebral Palsy After Robotic Assisted Gait Training Versus Body-Weight Supported Treadmill Training Objectives to Compare the Effect of Robotic-assisted Gait Training and Body-weight Supported Treadmill Training on Postural Stability in Ambulatory Children With Cerebral Palsy. Methods: A Randomized Control Study Involved Ambulatory Children With Cerebral Palsy With GMFCS Levels I, II and III. They Were Randomly Allocated to One of Two Locomotor Treadmill Training Groups. Postural Stability Outcomes Will Assessed Before and After the Intervention
Brief Title: Study Aims to Compare the Effect of Robotic-assisted Gait Training and Conventional Treadmill Training on Postural Stability in Ambulatory Children With Cerebral Palsy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Mozainah Yahya Aljoush, Clinical Specialist Physical Therapist working in Pediatric Outpatient Area in Physical Therapy Rehabilitation Department, at King Abdullah Specialized Children Hospital (KASCH), Ministry of National Guard Health Affair (MNGHA) Riyadh city Saudi Arabia, King Abdullah International Medical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KAIMRC study number RC19/363/R
Record Dates: First submitted 2024-11-20; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: CP (Cerebral Palsy); Robotic Exoskeleton; Treadmill Locomotor-based Training; Postural Stability
Keywords: Robotic Assited Gait Training; postural stability; CP
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robotic assisted gait training: participants in this group with receive gait training on the Lokomat (Active Comparator)
  Interventions: Device: Participants this group will receive gait training in robotic assisted gait training (RAGT) three times per week for eight weeks
- Body Weight Supported Treadmill Training: participants in this group receive training on Treadmill (Active Comparator)
  Interventions: Device: Body Weight Supported Treadmill Training

INTERVENTIONS:
Device: Participants this group will receive gait training in robotic assisted gait training (RAGT) three times per week for eight weeks — Robotic Assited Gait Training is a device used to train children with CP how to walk in effective manner by connecting their body to the harness, robotic devices that attached to the electronic treadmill
  Arms: Robotic assisted gait training: participants in this group with receive gait training on the Lokomat
Device: Body Weight Supported Treadmill Training — Participants in this group will receive gait training on conventional treadmill three times per week for eight weeks
  Arms: Body Weight Supported Treadmill Training: participants in this group receive training on Treadmill

SUMMARY:
The aim of this study is to explore the impact of gait training with a robotic device versus treadmill training on enhancing postural stability and walking capabilities in children with cerebral palsy (CP). The main questions to answer are children with CP who receive Robotic gait training will improve more in their postural stability compared with children with CP who received gait training on Treadmill? Are children with CP who receive Robotic gait training will improve more in their gross motor functions compared with children with CP who received gait training on Treadmill Are children with CP who receive Robotic gait training will improve more in their walking distance compared with children with CP who received gait training on Treadmill? Researchers will compare Group A to Group B to see if Robotic gait training has more effect on their outcomes than treadmill.

Participants will be randomly allocated to one of two group and will receive gait training for 3 times per week for eight weeks. Outcome measures will be assessed in the base line before starting intervention and after completing intervention.

Study Design A randomized control trial (RCT) Participants and Recruitment The trial will be conducted in Pediatric Out-Patient Rehabilitation Services (Clinic 750) at king Abdullah Specialized Children Hospital (KASCH), National Guard Hospital (NGH) in Riyadh, Saudi Arabia. The study populations are ambulatory children who have been diagnosed to have Spastic CP and who are referred and treated in rehabilitation department at KASCH in NGH in Riyadh. Recruitment will be through their medical record number. Inclusion Criteria are Spastic CP diagnosed from a pediatrician's (Neurology clinic) to have Diplegia, Hemiplegia, or Quadriparesis, Both gender with their age ranged from 5-14 years, independently able to stand and walk or walk with assistance, GMFCS Level I and II, with walking limitations, but able to ambulate without the gait device for most distances and with GMFCS Level III, who have a greater degree of walking limitation and able to use wheelchairs or walkers for short to long distances, Ability to follow instructions, Ability to accurately signal pain and discomfort using verbal or non-verbal signals, Ability to be participated in > 45 minutes of active Physical Therapy treatment, Hip's and knee's passive range of motion (ROM) within the minimum range requirement for robotic device (≤10° for hip and knee flexion contracture).

Exclusion Criteria are Botox injection in lower limb during the last 6 months, Surgical intervention in lower limb within a 1-year period prior to the examination date (including tendon release, muscle lengthening and bone surgery), Active drug for resisting epilepsy, Anatomical leg length differences larger than 2 cm (due to the limitations of robotic device), Bone-articular instability (joint dislocation), Fixed joint contractures; bone and joint deformities of lower extremities, Baclofen therapy by using an implanted infusion pump, Inhibiting casts for lower limb during 6 months prior to the program, Significant visual and hearing loss, Skin inflammation and open skin lesions around the lower limb or trunk, Any significant impairments in endurance due to limitation in cardiovascular system based on the patient's history, Cognition (higher mental functions) disorders resulted in lack of patient cooperation, Lack of consent from the parent or guardian.

Procedure We will send the invitation letter to the parents of participants. If interested, we will provide their parents with the informed consent (written). We will obtain the Assent from children who are unable to provide independent consent. Then, the participants will complete a basic screening session. If the participant met the eligibility criteria of the screening, he/ she will have a robotic device fitting assessment session to confirm there are no concerns with the participation in the study and to use the robotic device. If the participant met these the fitting criteria, the therapist would review the findings and will confirm (with the family) whether the child is eligible for the study based on their findings. The participants will be divided randomly to enter on of the two treatment groups (robotic or treadmill). Each participant will have a baseline assessment during the first two weeks prior to the beginning of the treatment, treatment program for eight weeks, and post treatment assessment at the last two weeks after completing the program. The duration of the whole program is twelve weeks. All participants will be assessed for their balance and walking parameters.

DETAILED DESCRIPTION:
Statement of problem:

Limitations in the literatures addressed the effect of robotic gait training on postural stability in CP children. Their limitation where varying levels of evidence, small sample size, different pediatric age groups with different functional levels, variation in setting program's frequency and duration of training and using a variety of assessment tools in assessing postural stability (Sarhan et al., 2014, Druzbicki et al., 2010, Druzbicki et al., 2013, Wallard et al., 2017). Lack of standardization in reporting of all aspects of the evaluation protocol for their assessment tools that used to measure postural stability such as; evaluation time, number of trials, arms and legs position at the time of assessment. This will lead to difficulty in replicating the study (Sarhan et al., 2014, Druzbicki et al., 2010, Druzbicki et al., 2013). The study compared between the effects of RAGT and BWSTT on postural stability did not address all aspects of static and dynamic postural stability. In addition, they did not report their standardization in their evaluation protocol (Sarhan et al., 2014). There was no study used CDP as a reliable, objective assessment tool with standardized protocols in assessing static and dynamic postural stability for CP children who are treated with RAGT compared to CP children who are treated with BWSTT. Since this assessment instrument can collaborate with the better understanding of all aspects concerning postural stability of children with CP, this study will fill the gaps in literature to guide future research that improves the postural control of children with CP.

Objectives of the study:

The primary objective of this study is to evaluate the comparative impact of RAGT and BWSTT for ambulatory children with CP on Static and Dynamic postural stability. The secondary objective is to evaluate the comparative impact of RAGT and BWSTT on Child's gross motor functions. The third objective is to evaluate the comparative impact of RAGT and BWSTT on Child's walking distance (endurance).

Hypothesis: Children with CP how are receiving the robotic gait training will not improve more on their postural stability compared with those receiving the BWSTT program.

Significance of the Study:

Reaching to the highest functional level, which is ambulation, is the main goal of children (and their care giver) with CP. Achieving this goal is vitally depending on improving their postural stability. RAGT holds promise for CP children in improving their postural stability that help in improving their ambulation functions. Both locomotor devices (treadmill and lokomat) provided walking training aiming to improve postural stability in CP patients. Robotic training device is expensive and not easy to be available in all clinics. It requires more time for preparing, adjusting, treating and removing the patient from the device, while the treadmill is accessible and available in most of the clinics, at also easy to administered and it require less time and effort from the therapist comparing to the robotic device. Measuring the comparative effects of both devices on postural stability will help us in rehabilitation clinical setting. If the study results show similar effects of both devices on postural stability, we will eliminate the effort and cost of ordering the expensive device (lokomat) and we will keep the cheaper device in our clinic (Treadmill). We can recommend robotic device to be used in other intensive rehabilitation setting as walking training aiming to improve gait related parameters. However, if the study results showed that; lokomat is superior to treadmill in improving postural stability; we will consider this in our future decision-making regarding requesting this expensive device.

Study Design:

A randomized control trial (RCT)

Participants and Recruitment:

The trial will be conducted in Pediatric Out-Patient Rehabilitation Services (Clinic 750) at king Abdullah Specialized Children Hospital (KASCH), National Guard Hospital (NGH) in Riyadh, Saudi Arabia. The study populations are ambulatory children who have been diagnosed to have Spastic CP and who are referred and treated in rehabilitation department at KASCH in NGH in Riyadh. Recruitment will be through their medical record number.

Inclusion Criteria:

1. Spastic CP diagnosed from a pediatrician's (Neurology clinic) to have Diaplegia, Diaparesis, Hemiplegia, Hemiparesis, or Quadriparesis.
2. Both gender with their age ranged from 5-14 years.
3. Independently able to stand and walk or walk with assistance.
4. GMFCS Level I and II, with walking limitations, but able to ambulate without the gait device for most distances and with GMFCS Level III, who have a greater degree of walking limitation and able to use wheelchairs or walkers for short to long distances.
5. Ability to follow instructions.
6. Ability to accurately signal pain and discomfort using verbal or non-verbal signals.
7. Ability to be participated in > 45 minutes of active Physical Therapy treatment.
8. Hip's and knee's passive range of motion (ROM) within the minimum range requirement for Lokomat (≤10° for hip and knee flexion contracture).

Exclusion Criteria:

1. Botox injection in lower limb during the last 6 months.
2. Surgical intervention in lower limb within a 1-year period prior to the examination date (including tendon release, muscle lengthening and bone surgery).
3. Active drug for resisting epilepsy.
4. Anatomical leg length differences larger than 2 cm (due to the limitations of Lokomat system).
5. Bone-articular instability (joint dislocation).
6. Fixed joint contractures; bone and joint deformities of lower extremities.
7. Baclofen therapy by using an implanted infusion pump.
8. Inhibiting casts for lower limb during 6 months prior to the program.
9. Significant visual and hearing loss.
10. Skin inflammation and open skin lesions around the lower limb or trunk.
11. Any significant impairments in endurance due to limitation in cardiovascular system based on the patient's history.
12. Cognition (higher mental functions) disorders resulted in lack of patient cooperation.
13. Lack of consent from the parent or guardian.

Sample size:

We will estimate the sample size based on the primary research question. The starting point for calculation of our sample size consideration is a one-group Locomotor study and using postural stability as the primary outcome. We will make the calculation by using the score of The Bruininks- Oseretsky Test of Motor Proficiency Subset 2 for balance baseline mean and standard deviation for one groups based on the study of Sarhan et al., (2014). Assuming the total mean difference in balance test of 1.8 and a pooled standard deviation of 1.7 units (Sarhan et al., 2014), the study will require a sample size of 15 participants for each group (i.e. a total sample size of 30, assuming equal group sizes), The desired power of the study will set at 80% and 5% significance level. We will increase the sample requirement to 36 to account for a potential drop out/ protocol deviation rate of 20%. The total sample size is 36 participants.

Ethical Consideration and Consent:

The current study will be approved by the Institutional Review Board (IRB) at King Saud University (KSU), Institutional Review Board (IRB) approval from king Abdullah International Medical Research Center (KAIMRC) in ministry of National Guard Health Affair (MNGHA) in Riyadh. Consent form will be completed by the parents and will be kept enclosed to ensure anonymity and Assent will be completed by children. Therapist is certified to use robotic training device (by having Lokomat user qualification Certificate in completion the training course on robotic rehabilitation therapy with the Lokomat).

Procedure:

We will send the invitation letter to the parents of participants. If interested, we will provide their parents with the informed consent (written). We will obtain the Assent from children who are unable to provide independent consent. Then, the participants will complete a basic screening session. If the participant met the eligibility criteria of the screening, he/ she will have a Lokomat fitting assessment session to confirm there are no concerns with the participation in the study and to use the Lokomat. If the participant met these the fitting criteria, the therapist will review the findings and will confirm (with the family) whether the child is eligible for the study based on their findings. The participants will be divided randomly to enter on of the two treatment groups (robotic or treadmill). Each participant will have a baseline assessment during the first two weeks prior to the beginning of the treatment, treatment program for eight weeks (Lunenburger et al., 2004), and post treatment assessment at the last two weeks after completing the program. The duration of the whole program is twelve weeks. All participants will be assessed for their balance and walking parameters.

Randomization:

Children who assigned a study ID number will attend their baseline assessment. Then, the child will be allocated to start at one of the two groups via a random assignment process by using a computer-generated random number system. The scheme of assignment will be prepared at the beginning of the study using a stratified randomization process (by using age and GMFCS level). At the end of the trial, this system will ensure that the number, age and GMFCS balance of participants who start in the robotic training group and treadmill training groups will be equal. A non-study research assistant (RA) will manage the randomization process through the entire study to allow blinding of the study investigators to the scheme, thus will eliminate the allocation bias.

Interventions:

Thirty sex participants will be divided randomly into two groups. The first group consists of 18 participants. They will receive robotic assisted gait training (RAGT) three times a week for four weeks for 45 minutes duration of session. The second group consists of 18 participants. They will receive body weight supported treadmill training (BWSTT) three times a week for four weeks for 45 minutes duration of session (Sarhan et al., 2014). Participants in both groups will receive a structural home-based individual physical therapy exercises program designed by physiotherapist. This program will mainly focus on stretching exercises, strengthening exercises and aerobic training for the main major muscles of upper and lower extremities (Fauzi et al., 2019). Exercises log will be provided to the participants. The duration of participation for each participant is approximately three months (twelve weeks) as folow; two weeks for baseline assessment, eight weeks for intervention period, and two weeks for post intervention assessment (Lunenburger et al., 2004). The follow-up for each participant during the study is three times per week (Sarhan et al., 2014).

Outcome Measures:

For the outcome measures, the evaluations will be performed twice; at the baseline (prior to the beginning of the treatment) and after finishing the treatment. The outcome measures will be assessed at single points in time to give the strength of objectivity of those outcome measures. The same examiner who will be blinded to the aims of the study and to which group the participant is allocated will perform all evaluation procedures.

The Primary Outcome Measure: Postural stability. The secondary Outcome Measure: gross motor functions. The third Outcome Measure: walking distance.

Statistical Analysis:

All statistical analyses will be performed with IBM SPSS Statistics (version 25) and datasets of all study participants will be analyzed on an intention-to-treat basis. Summary statistics (frequency, mean, standard deviation,) will be generated for all of the main demographic variables; gender, age, BMI, severity of CP according to GMFCS level, and treatment type. t- tests will be performed to determine statistically significant differences between the groups at baseline, statistically significant differences from pre- to post-training for each training group, and statistically significant differences between the training conditions on the outcomes: balance parameters, gross motor functions and Walking distance. Results will be presented as means ± standard deviation (SD) and the differences will be considered significant by keeping the Ninety-five percent confidence interval with a two-tailed level of significance set at p < 0.05 (Sarhan et al., 2014).

ELIGIBILITY:
Inclusion Criteria:

1. Spastic CP diagnosed from a pediatrician's (Neurology clinic) to have Diaplegia, Diaparesis, Hemiplegia, Hemiparesis, or Quadriparesis.
2. Both gender with their age ranged from 5-14 years.
3. Independently able to stand and walk or walk with assistance.
4. GMFCS Level I and II, with walking limitations, but able to ambulate without the gait device for most distances and with GMFCS Level III, who have a greater degree of walking limitation and able to use wheelchairs or walkers for short to long distances.
5. Ability to follow instructions.
6. Ability to accurately signal pain and discomfort using verbal or non-verbal signals.
7. Ability to be participated in > 45 minutes of active Physical Therapy treatment.
8. Hip's and knee's passive range of motion (ROM) within the minimum range requirement for Lokomat (≤10° for hip and knee flexion contracture).

Exclusion Criteria:

1. Botox injection in lower limb during the last 6 months.
2. Surgical intervention in lower limb within a 1-year period prior to the examination date (including tendon release, muscle lengthening and bone surgery).
3. Active drug for resisting epilepsy.
4. Anatomical leg length differences larger than 2 cm (due to the limitations of Lokomat system).
5. Bone-articular instability (joint dislocation).
6. Fixed joint contractures; bone and joint deformities of lower extremities.
7. Baclofen therapy by using an implanted infusion pump.
8. Inhibiting casts for lower limb during 6 months prior to the program.
9. Significant visual and hearing loss.
10. Skin inflammation and open skin lesions around the lower limb or trunk.
11. Any significant impairments in endurance due to limitation in cardiovascular system based on the patient's history.
12. Cognition (higher mental functions) disorders resulted in lack of patient cooperation.
13. Lack of consent from the parent or guardian.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2021-09-25 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Postural Stability using Computerized Dynamic Posturography (CDP) | Outcome measure performed at baseline (within 1-2 weeks before starting the intervention) and after ending the intervention (within 1-2 weeks after completing the intervention)

SECONDARY OUTCOMES:
Change in gross motor functions measured by GMFM-88 | Outcome measure performed at baseline (within 1-2 weeks before starting the intervention) and after ending the intervention (within 1-2 weeks after completing the intervention)

OTHER OUTCOMES:
Change in Walking Distance Measured by the 6-Minute Walk Test (6MWT) | Outcome measure performed at baseline (within 1-2 weeks before starting the intervention) and after ending the intervention (within 1-2 weeks after completing the intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Department, Physiotherapy Outpatient Clinic 750 at King Abdullah Specialized Children Hospital, Ministry of National Guard Health Affair, Riyadh, Saudi Arabia., Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aljosh M, Algabbani MF, Fagehi JM, Bawazeer M, Almohiza MA, Albishi AM, Alhusaini AA. Robotic versus treadmill training: Postural stability in ambulatory CP: RCT study. Pediatr Int. 2025 Jan-Dec;67(1):e70214. doi: 10.1111/ped.70214. PMID 41045011